CLINICAL TRIAL: NCT00437203
Title: Phase I Study of PF-00477736 With Gemcitabine In Patients With Advanced Solid Malignancies
Brief Title: PF-00477736 Is Being Studied In Advanced Solid Tumors In Combination With Chemotherapy With Gemcitabine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8211001
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasms
Keywords: Advanced cancer
MeSH Terms: conditions — Neoplasms | interventions — PF 00477736; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-00477736; Drug: gemcitabine

INTERVENTIONS:
Drug: PF-00477736 — * Escalating doses of PF-00477736 will be administered intravenously on Days 2 and 9 and gemcitabine will be administered intravenously on Days 1 and 8 of a 21-day cycle (doses to be evaluated range from 750 to 1250 mg/m2 in three separated cohorts).
  * If a patient is administered Cycle 0 - only PF-0047736 will be administered intravenously on Days 1 and 8 of a 21-day cycle for patients who have a 3-hour infusion and Days 1 and 8 of a 14-day cycle for patients who have a 24-hour infusion.
Drug: gemcitabine — gemcitabine will be administered intravenously on Days 1 and 8 of a 21-day cycle (doses to be evaluated range from 750 to 1250 mg/m2 in three separated cohorts).

SUMMARY:
To determine the overall safety of PF-00477736 when given in combination with gemcitabine, a chemotherapy agent, in patients with advanced solid tumors and determine the maximum dose of PF-00477736 that can be safely given in combination with gemcitabine. This is the first study of PF-00477736 in humans.

DETAILED DESCRIPTION:
The study was closed to enrollment as of 17 May 2010 due to business reasons. The patient on study continued treatment until 19 April 2011 when stopped for complete response. Premature closure was not prompted by any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytopathological diagnosis of solid malignancy that is refractory to standard therapy or for which no curative therapy exists.
* ECOG performance status 0 or 1.
* Adequate blood cell counts, kidney function and liver function.

Exclusion Criteria:

* Prior treatment with gemcitabine.
* Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
* NCI CTC Grade 2 or higher ARDS, non-infectious pneumonitis, or pulmonary fibrosis.
* NCI CTC Grade 2 or higher cardiovascular toxicities with the exception of NCI CTC Grade 3 hypertension that is well controlled.
* Known human immunodeficiency virus (HIV) seropositivity.
* Concurrent treatment with anticoagulants or known coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (3):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, New York, New York
- Pfizer Investigational Site, East Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1): PF-00477736 50 milligram (mg) 3 hours (hrs) infusion intravenously (IV) on Days 1 and 8 of cycle 0 and subsequently on Days 2 and 9 of each cycle (21 days cycle) for first 3 participants and on Days 2 and 9 of each cycle (21 days cycle), starting with cycle 1, for participants subsequently enrolled in this cohort. Gemcitabine 750 mg per square meter (mg/m^2) 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2): PF-00477736 65 mg 3 hrs infusion IV on Days 1 and 8 of cycle 0 and subsequently on Days 2 and 9 of each cycle (21 days cycle) for first 3 participants and on Days 2 and 9 of each cycle (21 days cycle), starting with cycle 1, for participants subsequently enrolled in this cohort. Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3): PF-00477736 80 mg 3 hrs infusion IV on Days 1 and 8 of cycle 0 and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4): PF-00477736 80 mg 24 hrs infusion IV on Days 1 and 8 of cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5): PF-00477736 120 mg 24 hrs infusion IV on Days 1 and 8 of cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6): PF-00477736 180 mg 24 hrs infusion IV on Days 1 and 8 of cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7): PF-00477736 270 mg 24 hrs infusion IV on Days 1 and 8 of cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle) for first 3 participants and on Days 2 and 9 of each cycle (21 days cycle), starting with cycle 1, for participants subsequently enrolled in this cohort. Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8): PF-00477736 340 mg 24 hrs infusion IV on Days 1 and 8 of cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine 750 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9): PF-00477736 infusion 180 mg 24 hrs infusion IV on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine infusion 1000 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle).
- PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10): PF-00477736 infusion 225 mg 24 hrs infusion IV on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine infusion 1000 mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle).
Period: Overall Study
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Started | 6 | 8 | 3 | 3 | 3 | 3 | 7 | 3 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 3 | 3 | 3 | 3 | 7 | 3 | 3 | 4
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Objective progression or relapse | 5 | 6 | 2 | 3 | 3 | 3 | 6 | 1 | 2 | 2
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1): PF-00477736 50 mg 3 hrs infusion IV on Days 1 and 8 of cycle 0 and subsequently on Days 2 and 9 of each cycle (21 days cycle) for first 3 participants and on Days 2 and 9 of each cycle (21 days cycle), starting with cycle 1, for participants subsequently enrolled in this cohort. Gemcitabine 750 mg mg/m^2 30 minutes infusion IV on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- Total: Total of all reporting groups
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10) | Total
Number analyzed (Participants) | 6 | 8 | 3 | 3 | 3 | 3 | 7 | 3 | 3 | 4 | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (18.3) | 62.3 (6.8) | 55.0 (5.2) | 45.0 (3.6) | 55.0 (11.5) | 44.3 (12.1) | 54.0 (8.9) | 55.7 (4.6) | 46.0 (6.9) | 49.5 (7.1) | 53.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 1 | 1 | 6 | 2 | 2 | 2 | 23
  Male | 4 | 6 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of PF-00477736 When Administered in Combination With Gemcitabine
Time Frame: Up to Day 21 Cycle 1
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg
Groups:
- PF-00477736 + Gemcitabine 750 mg/m^2: PF-00477736 infusion 50 mg, 65 mg or 80 mg IV administered over 3 hrs on Days 1 and 8 of Cycle 0 (21 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle), or PF-00477736 infusion 80 mg, 120 mg, 180 mg, 270 mg or 340 mg IV administered over 24 hrs on Days 1 and 8 of Cycle 0 (14 days cycle) and subsequently on Days 2 and 9 of each cycle (21 days cycle). Gemcitabine infusion 750 mg/m^2 IV administered over 30 minutes on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
- PF-00477736 + Gemcitabine 1000 mg/m^2: PF-00477736 infusion 180 mg or 225 mg IV administered over 24 hrs on Days 2 and 9 of each cycle (21 days cycle) along with gemcitabine infusion 1000 mg/m^2 IV administered over 30 minutes on Days 1 and 8 of each cycle (21 days cycle), starting with cycle 1.
Arm/Group | PF-00477736 + Gemcitabine 750 mg/m^2 | PF-00477736 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 36 | 7
mg | 270 | NA — MTD could not be determined as study was prematurely terminated.

2. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: OR based assessment of confirmed complete response(CR)/confirmed partial response(PR)/stable disease(SD)/progressive disease(PD) as per Response Evaluation Criteria in Solid Tumors(RECIST).CR:disappearance of target lesions;PR:at least(>=) 30% decrease in sum of longest dimensions of target lesions(reference:baseline sum of longest dimensions);PD:>=20% increase in sum of longest dimensions of target lesions(reference:smallest sum of longest dimensions recorded since treatment started)/appearance of any new lesions;SD:no adequate shrinkage to qualify for PR/adequate increase to qualify for PD.
Time Frame: Baseline, Day 15 of Cycle 2 and 4 and every 4 cycles thereafter up to Week 62
Population: FAS included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 6 | 8 | 3 | 3 | 3 | 3 | 7 | 3 | 3 | 4
participants | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0(pre-dose), 0.25, 1, 3, 3.25, 3.5, 4, 6, 8, 10, 24 hr post-infusion start:Day 1, 8 Cycle 0 Cohort 1-3; 0(pre-dose), 0.25, 1, 2, 24, 24.25, 24.5, 25, 27, 29, 31, 48 hr post-infusion start:Day 1-2, 8-9 Cycle 0 Cohort 4-8; Day 2-3, 9-10 Cycle 1 Cohort 9-10
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)]
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: 0(pre-dose), 0.25, 1, 3, 3.25, 3.5, 4, 6, 8, 10, 24 hr post-infusion start: Day 1, 8 Cycle 0
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-48)]
Description: AUC (0-48)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-48).
Time Frame: 0(pre-dose), 0.25, 1, 2, 24, 24.25, 24.5, 25, 27, 29, 31, 48 hr post-infusion start:Day 1-2, 8-9 Cycle 0 Cohort 4-8; Day 2-3, 9-10 Cycle 1 Cohort 9-10
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Concentration of PF-00477736 in Urine
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Metabolite Profile of PF-00477736 in Plasma and Urine
Time Frame: as for outcome 3
Population: Data was not analyzed, as study was terminated due to business reasons.
Measure: Number; unit: percentage of recovered metabolite
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10)
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/8 | 2/3 | 1/3 | 0/3 | 2/3 | 4/7 | 2/3 | 0/3 | 3/4
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 3/3 | 3/3 | 3/3 | 3/3 | 7/7 | 2/3 | 3/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) (N=6) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) (N=8) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) (N=3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) (N=3) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) (N=3) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) (N=3) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) (N=7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) (N=3) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) (N=3) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10) (N=4)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venoocclusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00477736 50 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 1) (N=6) | PF-00477736 65 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 2) (N=8) | PF-00477736 80 mg 3 Hrs + Gemcitabine 750 mg/m^2 (Cohort 3) (N=3) | PF-00477736 80 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 4) (N=3) | PF-00477736 120 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 5) (N=3) | PF-00477736 180 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 6) (N=3) | PF-00477736 270 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 7) (N=7) | PF-00477736 340 mg 24 Hrs + Gemcitabine 750 mg/m^2 (Cohort 8) (N=3) | PF-00477736 180 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (Cohort 9) (N=3) | PF-00477736 225 mg 24 Hrs + Gemcitabine 1000 mg/m^2 (cohort10) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 3 | 1 | 1 | 5 | 1 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 2 | 1 | 1 | 1 | 3 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 1 | 2 | 2 | 4 | 1 | 3 | 1
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 2 | 0
Catheter site discharge (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 7 | 3 | 2 | 1 | 1 | 5 | 1 | 3 | 1
Infusion site erythema (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 4 | 1 | 3 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin graft infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.